CLINICAL TRIAL: NCT02128425
Title: Phase II Randomized Controlled Trial of FOLFOXIRI Compared to FOLFOX in First Line Treatment of Chemo-naive Metastatic Colorectal Cancer
Brief Title: FOLFOXIRI Compared to FOLFOX in First Line Treatment of Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, M.D, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GIHSYSU06
Record Dates: First submitted 2014-04-15; First posted 2014-05-01 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-04

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Colorectal cancer; Metastatic colorectal cancer; FOLFOXIRI; FOLFOX; Oxaliplatin; irinotecan; Leucovorin; 5-FU
MeSH Terms: conditions — Colorectal Neoplasms | interventions — FOLFOXIRI protocol; Irinotecan; Oxaliplatin; Leucovorin; Fluorouracil; Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FOLFOXIRI (Experimental): FOLFOXIRI
  Interventions: Drug: FOLFOXIRI
- FOLFOX (Active Comparator): FOLFOX
  Interventions: Drug: FOLFOX

INTERVENTIONS:
Drug: FOLFOXIRI — irinotecan* 165 mg/m² + oxaliplatin 85 mg/m² + leucovorin 200 mg/m² + 5-FU 3200 mg/m² cont. inf. 46h all on day 1 of each 2 weeks cycle
  *reduced in UGT1A1 7/7 patients
  Other Names: Irinotecan; Oxaliplatin; Leucovorin; 5-Fluorouracil
  Arms: FOLFOXIRI
Drug: FOLFOX — oxaliplatin 85 mg/m² + leucovorin 400 mg/m² +5-FU 400mg/m² bolus iv.+ 5-FU 2400 mg/m² cont. inf. 46h all on day 1 of each 2 weeks cycle
  Other Names: Oxaliplatin; Leucovorin; 5-Fluorouracil
  Arms: FOLFOX

SUMMARY:
The purpose of the study is to evaluate if the exposure to all the three active cytotoxic agents (FOLFOXIRI regimen) is superior in terms of progression-free survival to conventional chemotherapy with the FOLFOX regimen as first-line treatment of chemo-naive metastatic colorectal cancer patients.

A second primary aim is to evaluate the response rate, safety and tolerability of the chemotherapy of FOLFOXIRI regimen in this patient population.

Patients will be randomized to two therapy groups:

Experimental arm A: Chemotherapy with FOLFOXIRI Standard arm B: Chemotherapy with FOLFOX

DETAILED DESCRIPTION:
Survival of patients with metastatic colorectal cancer is correlated with the proportion of patients who receive all the three active drugs , but not with the proportion of patients who receive any second-line therapy. A superior efficacy in PFS,ORR and OS of FOLFOXIRI has been reported with acceptable toxicity. Moreover,evidence suggests that continuous dosing metronomic chemotherapy may be more efficacious than interval-chemotherapy.

Therefore, a way to improve the outcome of metastatic colorectal cancer patients could be to administer a maintenance first-line regimen containing the three active agents.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained before any study specific procedures. -Subjects must be able to understand and willing to sign a written informed consent.
* Male or female subjects ≥ 18 years ≤ 75 years of age
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 2.(ECOG PS 0-2 for≥18 years ≤ 65 years of age ，ECOG PS 0-1 for >65 years of age)
* Histological or cytological documentation of adenocarcinoma of the colon or rectum. All other histological types are excluded.
* There must be documentation by PET/CT scan, CT scan, MRI, or intraoperative palpation (at the time of resection of the primary colorectal tumor, if applicable) that the patient has evidence of metastases (Histologic confirmation of metastasis is not required.).
* At least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria measured within 4 weeks prior to registration.
* No previous chemotherapy or target therapy for metastatic disease (adjuvant chemotherapy for non-metastatic disease is allowed if terminated more than 6 months ago).
* In case of previous radiotherapy, at least one measurable lesion should be located outside the irradiated field.
* Adequate bone marrow, hepatic and renal function as assessed by the following laboratory requirements conducted within 7 days of starting study treatment:
* Leukocytes ≥ 3.0 x109/ L, absolute neutrophil count (ANC) ≥ 1.5 x109/ L, platelet count ≥ 100 x109/ L, hemoglobin (Hb) ≥9g/ dL.
* Total bilirubin ≤ 1.5 x the upper limit of normal (ULN).
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5 x ULN.
* Alkaline phosphatase limit ≤ 5x ULN.
* Amylase and lipase ≤ 1.5 x the ULN.
* Serum creatinine ≤ 1.5 x the ULN.
* Calculated creatinine clearance or 24 hour creatinine clearance ≥ 50 mL/ min.

Exclusion Criteria:

* Previous palliative chemotherapy for metastatic disease，previous adjuvant chemotherapy including irinotecan or oxaliplatin within 6 months before random assignment.
* Previous or concurrent cancer that is distinct in primary site or histology from colorectal cancer within 5 years prior to randomization.
* Life expectancy > 12 weeks;
* Extended field radiotherapy within 4 weeks or limited field radiotherapy within 2 weeks prior to randomization. Subjects must have recovered from all therapy-related toxicities.
* Major surgical procedure, open biopsy, or significant traumatic injury within 4 weeks before start of study medication.
* Congestive heart failure ≤ New York Heart Association (NYHA) class 2.
* Significant cardiovascular disease including unstable angina or myocardial infarction within 6 months before initiating study treatment or a history of ventricular arrhythmia
* Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within the 6 months before start of study medication.
* Any evidence of active infection.
* History of interstitial pneumonitis or pulmonary fibrosis
* Pregnancy or lactation at the time of study entry.
* Known dihydropyrimidine dehydrogenase (DPD) deficiency
* Any illness or medical conditions that are unstable or could jeopardize the safety of the subjects and his/her compliance in the study.
* Active inflammatory bowel disease or other bowel disease causing chronic diarrhoea
* Subjects with known allergy to the study drugs or to any of its excipients.
* Current or recent (within 4 weeks prior to starting study treatment) treatment of another investigational drug or participation in another investigational study.
* Continuous use of immunosuppressive agents (except the use of corticosteroids as anti-emetic prophylaxis/treatment).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2014-04; Primary Completion 2017-02 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival after induction and maintenance chemotherapy (PFS1) | up to 18 months
  Progressions are evaluated every 8 weeks according to WHO criteria and reviewed by an independent panel at the end of follow up (36 months).

SECONDARY OUTCOMES:
Progression-free survival after re-introduction of chemotherapy (PFS2) | up to 24 months
Response rate during re-introduction of chemotherapy | up to 12 months
  (CR + PR rate according to RECIST)
Early tumor shrinkage rate in 8 weeks after induction treatment | 8 weeks
Overall survival | up to 5 years
toxicity and safety | up to 24 months
  Number of participants with adverse events as a measure of safety and tolerability according to NCI CTC 4.0
QLQ (QLQ C30) - scores according to EORTC QLQ-C30 scoring manual (Quality of life) | up to 36 months
Translational research | up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Yanhong Deng, M.D., Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- Gastrointestinal Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China